CLINICAL TRIAL: NCT04040543
Title: Development of a Biomarker to Assess Adherence to Nutrients Supplements
Brief Title: Development of a Marker of Adherence for Tracking Consumption of Nutrient Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1410234
Record Dates: First submitted 2019-07-24; First posted 2019-07-31 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Adherence, Treatment
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Daily (Experimental): Daily supplementation with product containing markers
  Interventions: Dietary Supplement: lipid-based nutrient supplement containing adherence markers
- Intermittent (Experimental): Daily supplementation with either the product containing markers or the product not containing markers
  Interventions: Dietary Supplement: lipid-based nutrient supplement containing or not containing adherence markers
- Control (Placebo Comparator): Daily supplementation with product not containing markers
  Interventions: Dietary Supplement: lipid-based nutrient supplement not containing adherence markers

INTERVENTIONS:
Dietary Supplement: lipid-based nutrient supplement containing adherence markers — The supplement will be provided once daily for 10 days
  Arms: Daily
Dietary Supplement: lipid-based nutrient supplement containing or not containing adherence markers — The product containing adherence markers will be provided once daily every other day (5 days total); the product not containing adherence markers will be provided on the intervening days for a total of 10 days.
  Arms: Intermittent
Dietary Supplement: lipid-based nutrient supplement not containing adherence markers — The supplement will be provided once daily for 10 days
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether selected adherence markers can be used to track daily or intermittent consumption of nutrient supplements.

DETAILED DESCRIPTION:
The investigators will assess whether urinary concentrations of selected adherence markers can be used to distinguish between daily or intermittent consumption of lipid-based nutrient supplements.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant, non-lactating women

Exclusion Criteria:

* BMI <18.5kg/m2 or >25.0 kg/m2
* Diagnosis of chronic disease
* Use of medication that can affect gastrointestinal mobility
* Consumption of more than 7 alcoholic drinks per week
* Smoking
* Unwillingness to refrain from consuming dietary sources of the marker compound(s) 3 days prior to, and during the 12 day urine collection period
* Unwillingness to adhere to the study protocol
* Peanut allergy
* Cow milk allergy
* Soy allergy
* Almond allergy
* Allergy to adherence markers
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
urinary concentration of saccharin (nmol/L) | change in concentration between study day 4 (baseline) and study days 7,8,12,13 and 15
urinary concentration of saccharin (nmol/g creatinine) | change in concentration between study day 4 (baseline) and study days 7,8,12,13 and 15
urinary concentration of resveratrol metabolites (nmol/L) | change in concentration between study day 4 (baseline) and study days 7,8,12,13 and 15
  resveratrol metabolites may include resveratrol glucuronides and/or resveratrol sulfates
urinary concentration of resveratrol metabolites (nmol/g creatnine) | change in concentration between study day 4 (baseline) and study days 7,8,12,13 and 15
  resveratrol metabolites may include resveratrol glucuronides and/or resveratrol sulfates

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Haskell, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States